CLINICAL TRIAL: NCT01780077
Title: A Phase 1 Single Center, Randomized, Double-Blind, Ascending, Multi-Dose, Within-Subject Controlled Study of RXI-109 for the Treatment of Incision Scars Made in the Abdominal Skin of Healthy Subjects
Brief Title: Evaluation of Safety, PK, and Preliminary Effects on Scar Formation of Multiple Intradermal Administrations of RXI-109
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: RXi Pharmaceuticals, Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: RXI-109-1202
Record Dates: First submitted 2013-01-28; First posted 2013-01-30 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Cicatrix; Scar Prevention
Keywords: Scar; Scar prevention; Fibrosis
MeSH Terms: conditions — Cicatrix; Fibrosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RXI-109 (Experimental)
  Interventions: Drug: RXI-109; Drug: Placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: RXI-109; Drug: Placebo

INTERVENTIONS:
Drug: RXI-109 — Multiple intradermal injections of RXI-109 at incision sites
Drug: Placebo — Multiple intradermal injections of placebo at incision sites

SUMMARY:
The purpose of this trial is to evaluate the safety and tolerability of multiple (3) intradermal doses of RXI-109 at small surgical incisions in the abdominal skin of healthy volunteers. The effect of RXI-109 versus placebo on scarring at these incision sites will be evaluated visually, histologically, and by biomarker analysis.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 21-50 years of age
* General good health; if female not pregnant or lactating
* Phototype 3 and above based on the Fitzpatrick scale.

Exclusion Criteria:

* Pregnant or lactating
* Use of tobacco or nicotine-containing products within 1 month prior to enrollment and while on study
* Type 1 or 2 diabetes mellitus
* A history or presence of any medical condition or therapy that would make the subject an unsafe candidate in the opinion of the investigator

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2012-12; Primary Completion 2014-06 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of multiple intradermal administrations of RXI-109 | 12 weeks
  Evaluate safety and tolerability of multiple administrations of RXI-109 at the site of intradermal injection. Examine and assess any and all local and systemic toxicities

SECONDARY OUTCOMES:
To assess the effect of multiple intradermal administrations of RXI-109 on scar formation | 12 weeks
  Assess visual outcome and histology of scars. Digital images of the RXI-109 and placebo-treated incisions/scars will be captured and scored.

OTHER OUTCOMES:
To assess the timeline and levels of biomarkers | 12 weeks
  Analysis of immunohistochemical analysis of biomarkers common to the scar formation pathway.